CLINICAL TRIAL: NCT05182749
Title: A Phase 1/2a Double-Blind, Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of Oral Administration of the Bacteriophage Preparation, ShigActive™, in a Human Experimental Model of Shigellosis With Shigella Flexneri 2a Strain
Brief Title: Safety and Efficacy of the Bacteriophage Preparation, ShigActive™, in a Human Experimental Model of Shigellosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intralytix, Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITX/SA-001; Shigella CVD 32000 (Other: Center for Vaccine Development & Global Health); HP-00097063 (Other: University of Maryland, Baltimore)
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Shigellosis
Keywords: bacteriophage; phage; Shigella
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dose is 1mL of placebo given orally three times a day for 7 days (Phase 1) or 6 days (Phase 2a)
  Interventions: Other: Placebo
- Bacteriophage (Experimental): Dose is 1mL of bacteriophage preparation given orally three times a day for 7 days (Phase 1) or 6 days (Phase 2a)
  Interventions: Biological: bacteriophage

INTERVENTIONS:
Biological: bacteriophage — A cocktail of lytic Shigella-specific bacteriophages orally administered with sodium bicarbonate solution
  Other Names: ShigActive
  Arms: Bacteriophage
Other: Placebo — Placebo orally administered with sodium bicarbonate solution
  Other Names: Phosphate Buffered Saline
  Arms: Placebo

SUMMARY:
The study is a first-in-human Phase 1/2a randomized, double-blind, placebo-controlled trial to assess the clinical safety and efficacy of ShigActive in healthy adults with experimental Shigella challenge.

DETAILED DESCRIPTION:
The purpose of this study is to determine if ShigActive is safe and effective in healthy adults in a continuous Phase 1/2a trial. Phase 1 will asses the safety of ShigActive in healthy adults, while Phase 2a will evaluate the safety and efficacy of ShigActive in healthy adults after a challenge with Shigella.

ShigActive is a collection of bacteriophages. Bacteriophages (or phages) are viruses that infect only bacteria. The phages in ShigActive infect a specific type of bacteria called Shigella, which is the causative agent of shigellosis or dysentery. ShigActive is intended to significantly reduce or eliminate Shigella levels in the human gastrointestinal tract, which in turn, is anticipated to reduce the incidence and/or severity of shigellosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years.
2. Access to CVD clinical site and available and willing to be followed for the planned duration of the study, including all follow-up visits.
3. Able and willing to provide informed consent.
4. Willing to participate after all aspects of trial explained.
5. Assessment of understanding:

   1. Volunteer demonstrates understanding of this study;
   2. Completes a questionnaire prior to first treatment with verbal demonstration of understanding of all questionnaire items answered incorrectly;
   3. Receives a passing score of 70% or higher on the Comprehension Assessment Tool.
6. Agrees not to enroll in another study of an investigational research agent during the study, with the exception of potentially life-saving or COVID-19-related experimental treatments.
7. Good general health as shown by medical history, physical exam, and screening laboratory tests or clinical laboratory abnormalities per clinical judgment of the PI.
8. Agrees not to donate blood or blood products during participation in the study or for 30 days after completion of study participation.
9. Within normal/acceptable laboratory ranges during screening including:

   1. Absolute neutrophil count (1,500-8,000/mm^3; 1,200-8,000/mm^3 for African-American subjects);
   2. Bilirubin (<1.4 mg/dL unless known Gilbert's syndrome, then >2.0 mg/dL);
   3. Serum IgA (≥70 mg/dL or below lower limit of normal range);
   4. HLA-B27 negative (Phase 2a only);
   5. Stool culture (No Salmonella, Shigella, Campylobacter, Yersinia; presence of normal flora; no pathogenic protozoa by microscopic examination).
10. Hemoglobin ≥11.5 g/dL for volunteers who were assigned female sex at birth, ≥13.0 g/dL for volunteers who were assigned male sex at birth.

    a. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (i.e., a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
11. White blood cell count = 3,300 to 11,000 (2,800-11,000 for African-Americans) cells/mm^3.
12. Total lymphocyte count ≥800 cells/mm^3.
13. Remaining differential either within institutional normal range or with site physician approval.
14. Platelets = 125,000 to 450,000/mm^3.
15. Chemistry panel: alanine aminotransferase (ALT) <1.25 times the institutional upper limit of normal and creatinine ≤ institutional upper limits of normal.
16. Negative HIV-1 and -2 blood test: must have a negative FDA-approved enzyme immunoassay (EIA).
17. Negative for HBsAg.
18. Negative for HCV antibody.
19. Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to enrollment and within 24 hours of initial treatment.

    a. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy are not required to undergo pregnancy testing.
20. Reproductive status: A volunteer who was assigned female sex at birth must agree to use adequate contraception, defined as consistent and correct use of an FDA-recommended contraceptive method or combination of methods in accordance with the product label. For example:

    1. Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide, and another method such as prescription hormonal contraceptive;
    2. Intrauterine device (IUD);
    3. Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch) subdermal, or intramuscular route used in combination with another method, such as barrier methods;
    4. Total abstinence;
    5. Sterilization of a female participant's monogamous male partner prior to entry into the study;
    6. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation.
21. Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.
22. Phase 2a only: Available for a 12-day inpatient stay.
23. Phase 2a only: Fully vaccinated against COVID-19 for at least 30 days prior to enrollment.
24. Phase 2a only: Successful completion of inpatient acclimation period on Day -1.

Exclusion Criteria:

1. Blood products received within 120 days before first treatment.
2. Investigational research agents received within 30 days before first treatment.
3. Body mass index (BMI) less than 19.0 kg/m2 or greater than 36.0 kg/m2.
4. Pregnant or breastfeeding.
5. Poor venous access, as defined by inability to obtain venous blood after 3 venipuncture attempts.
6. Persons whose occupation involves the handling of ETEC, cholera, or Shigella bacteria.
7. Regular (one time per week or more) use of antidiarrheals, stool softeners, laxatives, antacids, or other agents to lower stomach acidity.
8. Use of oral or IV antimicrobials within 2 weeks of study start or planned use during active study phase.
9. Proton pump inhibitors, H2 blockers or antacids within 48 hours prior to dosing or planned use during active study phase.
10. Abnormal bowel patterns, defined by <3 stools per week or >2 stools per day on average over the past 6 months.
11. Taking supplemental probiotics in the form of pills or tablets within 2 weeks of enrollment or during study period.
12. Received prior vaccines, challenges or known exposure to (e.g., laboratory worker) Shigella within the past 3 years.
13. Live attenuated vaccines received within 30 days before first study treatment or scheduled within 14 days after the first study treatment (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine).
14. Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first treatment (e.g., COVID-19, tetanus, pneumococcal, hepatitis A or B).
15. Allergy treatment with antigen injections within 30 days before first treatment or that are scheduled within 14 days after first treatment.
16. Immunosuppression as the result of an underlying illness
17. Immunosuppressive medications received within 30 days before first treatment or planned use during study (Not exclusionary: 1) corticosteroid nasal spray; 2) inhaled corticosteroids; 3) topical corticosteroids for mild, uncomplicated dermatitis; or 4) a single course of oral/parenteral prednisone or equivalent at doses <60 mg/day and length of therapy <11 days with completion at least 30 days prior to enrollment).
18. Immunoglobulin received within 60 days before first treatment.
19. Autoimmune disease (Not exclusionary: mild, well-controlled psoriasis).
20. History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up.)
21. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    1. A process that would affect the immune response;
    2. A process that would require medication that affects the immune response;
    3. Any contraindication to repeated injections or blood draws;
    4. A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period;
    5. A condition or process for which signs or symptoms could be confused with reactions to treatment or challenge;
    6. Any condition specifically listed among the exclusion criteria below:

       • Chronic liver disease, renal insufficiency, unstable or progressive neurological disorders, diabetes mellitus, collagen vascular disease (such as lupus), active neoplastic disease (not cured or in remission), previous hematological malignancy, or seizure since the age of 21 years;
    7. Any of the following in the past 10 years: Crohn's disease, ulcerative colitis, irritable bowel disease, celiac disease, stomach or intestinal ulcers, or 2 or more episodes of inflammatory arthritis (joint pain and swelling);
    8. Any history of recurrent infections;
    9. Any current illness requiring daily medication (vitamins, birth control pills, nasal or topical medications, allowed);
    10. Blood in stool on >2 occasions (other than small amounts from straining) in past 12 months;
    11. Recurrent diarrhea (>5 episodes in past 6 months, each lasting >3 days or more).
22. History of excessive alcohol consumption or drug dependence within last 3 years
23. Any medical, psychiatric, occupational, or other condition that, in the judgment of the Investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
24. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions.)
25. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the Investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study.)
26. Seizure disorder/epilepsy: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years
27. Asplenia: any condition resulting in the absence of a functional spleen
28. History of chronic GI illness, including severe dyspepsia, lactose intolerance, or other significant GI tract disease (e.g., irritable bowel syndrome, inflammatory bowel syndrome, gastric ulcer disease)
29. Any other criteria which, in the Investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study
30. Phase 2a only: Occupation as a food handler, in child-care, in elder-care or as a healthcare worker with direct contact from challenge to 4 weeks after discharge home.
31. Phase 2a only: Serum Shigella flexneri 2a LPS IgG titer of ≥2500
32. Phase 2a only: History of diarrhea in the 7 days prior to treatment (outpatient diarrhea is defined as ≥ 3 unformed [Grade 3 or greater] loose stools in 24 hours).
33. Phase 2a only: Screening stool culture positive for the presence of Salmonella, Shigella, Campylobacter, Yersinia, Vibrio cholera or presence of pathogenic protozoa by microscopic examination.
34. Phase 2a only: Screening stool culture with an absence of normal flora.
35. Phase 2a only: Subjects who are unwilling to abstain from taking antipyretics or analgesics during the 7 days following treatment.
36. Phase 2a only: Persons with IgA deficiency (serum IgA <70 mg/dL)
37. Phase 2a only: Symptoms of traveler's diarrhea associated with travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within 3 years prior to dosing
38. Phase 2a only: History of shigellosis within the last 3 years
39. Phase 2a only: History of the following types of abdominal surgery:

    1. Any major GI surgery (e.g., intestinal resection or splenectomy);
    2. Laparoscopic abdominal surgery within the past year;
    3. Presence of a large abdominal scar of unclear origin.
40. Phase 2a only: Known significant allergy to ciprofloxacin or trimethoprim-sulfamethoxazole.
41. Phase 2a only: Electrocardiogram (ECG) with clinically significant findings or features that would interfere with the assessment of myo/pericarditis, as determined by a contract ECG Lab or cardiologist, including any of the following:

    1. Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS ≥120 ms, PR interval ≥220 ms, any second or third degree AV block, or QTc prolongation >450 ms);
    2. Repolarization (ST segment or T wave) abnormality that will interfere with the assessment of myo/pericarditis;
    3. Significant atrial or ventricular arrhythmia;
    4. Frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, 2 premature ventricular contractions in a row);
    5. ST elevation consistent with ischemia;
    6. Evidence of past or evolving myocardial infarction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number and Severity of Solicited and Unsolicited Adverse Reactions | Up to Day 90
  Number of subjects reporting solicited and unsolicited AEs, laboratory measures of safety, and adverse (up to Day 29) and serious adverse events (up to Day 90) following treatment with ShigActive or placebo
Phase 2a: Onset of Clinical Shigellosis Post-Challenge | Day 2 to Day 7 (Post-Challenge)
  Clinical shigellosis with onset during Day 2 to Day 7 post-challenge, defined as fever, diarrhea, and/or dysentery
Phase 2a: Number of Solicited and Unsolicited Adverse Reactions | Up to Day 90
  Number of subjects reporting solicited and unsolicited AEs, laboratory measures of safety, and adverse (up to Day 29) and serious adverse events (up to Day 90) following treatment with ShigActive or placebo

SECONDARY OUTCOMES:
Phase 2a: Onset of Moderate-to-Severe Shigellosis Post-Challenge | Day 2 to Day 7 (Post-Challenge)
  Moderate-to-severe shigellosis with onset during Day 2 to Day 7 post-challenge, defined using graded disease severity scoring methods (Grade 3 [mild] to Grade 5 [severe]) defined by number of loose stools, fever, dysentery, and abdominal cramping
Phase 2a: Severity of Shigellosis Symptoms | Day 2 to Day 7 (Post-Challenge)
  Severity of shigellosis symptoms (e.g., diarrhea, dysentery, fever) using graded severity scoring methods (Grade 1 [mild] to Grade 3 [severe])
Phase 2a: Number of Shigella Organisms Secreted in Stool | Up to Day 15
  Qualitative and quantitative (mean, median and geometric mean colony forming units [CFUs]) assessment of Shigella challenge strain shedding in stool samples following treatment with ShigActive or placebo, and challenge with Shigella

OTHER OUTCOMES:
Phase 1: Effect on Gut Microbiome Community States | Up to Day 29
  Assess the effect of oral phage administration on the gut microbiome in stool samples following treatment with ShigActive or placebo using next generation sequencing
Phase 1: Number of Shigella-specific Bacteriophage Shed in Stool | Up to Day 29
  Quantitation (mean, median and geometric mean plaque forming units [PFUs]) of bacteriophage shedding in stool samples following treatment with ShigActive or placebo
Phase 2a: Number of Shigella-specific Bacteriophage Shed in Stool | Up to Day 15
  Quantitation (mean, median and geometric mean PFUs) of bacteriophage shedding in stool samples following treatment with ShigActive or placebo
Phase 2a: Geometric Mean Anti-Shigella Antibody Titers | Up to Day 90
  Magnitude of response (geometric mean titer [GMT] and geometric mean peak titer) of fecal and serum IgA and IgG antibodies to LPS and Ipas following treatment with ShigActive or placebo and challenge with Shigella
Phase 2a: Geometric Mean anti-LPS Antibody Secreting Cell (ASC) Responses | Up to Day 8
  Quantitation (point estimate, 95% confidence interval [CI], mean, median and geometric mean) of IgG anti-LPS ASC responses in circulating peripheral blood mononuclear cells (PBMCs) following treatment with ShigActive or placebo, and challenge with Shigella

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sulakvelidze, PhD, Study Director — Intralytix, Inc.; Wilbur Chen Chen, MD, MS, Principal Investigator — University of Maryland, Baltimore, Center for Vaccine Development and Global Health
Locations (1):
- University of Maryland, Baltimore, University of Maryland School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No